CLINICAL TRIAL: NCT02312778
Title: Immediate Effects of a Spinal Lumbar Manipulation on the Threshold Pressure Pain and the Postural Control in Subjects With Non-specific Low Back Pain
Brief Title: Immediate Effects of a Spinal Lumbar Manipulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Jefferson Fagundes Loss, Professor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AVBA x COP
Record Dates: First submitted 2014-11-28; First posted 2014-12-09 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Low Back Pain
Keywords: non-specific low back pain; center of pressure; spinal lumbar manipulation; high velocity and low amplitude manipulation; postural control
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- HVLA Manipulation (Experimental): Intervention Group who receives a high velocity and low amplitude (HVLA) lumbar manipulation. A manual procedure also known as high velocity and low amplitude lumbar spinal manipulation is delivered to the subjects in the side lying position. The more restricted lumbar segment (mobility restriction) will be the target region for the manipulative procedure.
  Interventions: Other: HVLA Manipulation
- Sham Manipulation (No Intervention): Control Group who receives a simulated manipulation.

INTERVENTIONS:
Other: HVLA Manipulation — Intervention Group who receives a high velocity and low amplitude (HVLA) lumbar manipulation. A manual procedure also known as high velocity and low amplitude lumbar spinal manipulation are delivered for the subjects in the side lying position. The lumbar segment more restrict (mobility restriction) will be the target region for the manipulative procedure.
  Arms: HVLA Manipulation

SUMMARY:
Non-specific low back pain is defined as a pain with no specific vertebral-related cause, such as infectious disease, tumor, osteoporosis, fracture, structural abnormality, inflammatory disease, radicular compressive syndrome or cauda equine syndrome. Non-specific low back pain is a common disease in many countries. This musculoskeletal disorder is costly to public health systems. Therefore, the use of manual therapies is important in the treatment of this disease and studies show the effectiveness of this type of therapy.

Spinal manipulation is applied in manual therapies such as Osteopathy, Chiropractic and Physical Therapy and is widely used for acute and chronic non-specific low-back pain. There is moderate evidence that spinal manipulation is superior to sham spinal manipulation for improving short-term pain and function in chronic and acute non-specific low back pain. However the therapeutic mechanisms involved in this procedure are not well understood. Furthermore, while the high velocity and low amplitude spinal therapy has been shown to be effective in reducing pain and improving functional capacity in subjects with non-specific low back pain, the effect on postural variables have not been investigated. Therefore, the aim of this study is to evaluate the acute effect of lumbar manipulation on pain and postural variables.

Twenty-four individuals with non-specific low back pain will be randomly allocated to two groups. The intervention group will receive high velocity and low amplitude spinal therapy, while the control group will receive sham manipulation. Immediately before and after the respective manipulation protocol, both groups will be evaluated regarding pain level, using a visual-analogue scale and algometer, and postural variables, using center of pressure displacement measured with the aid of a force plate. While the patient and therapist manipulator will be aware of the protocol applied in each case, the evaluator will be blind. A statistical treatment will be used to compare the results.

DETAILED DESCRIPTION:
Mean and standard deviation are calculated for each variable of postural control, as well as the values obtained in the measurement of pain using the numeric pain rating scale and algometry data.

t-test or Mann-Whitney test will be used to compare data before and after the manipulation protocol.

Multiple One-Way ANOVAs will be used to compare the manipulation protocol, for each dependent variable: effects of pain and center of pressure displacement.. Statistical analysis will be conducted with a confidence interval of 95%, α value of 5%, p value of ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* recurrent low back pain in the last three months;
* medical diagnosis of non-specific low back pain, daily or almost daily;
* subjects that will present at least four variables which encompass the clinical prediction rule: symptoms duration less than 16 days, Fear Avoidance-Beliefs Questionnaire score lower than 19 in the work subscale, segmental lumbar hypermobility test in prone decubitus, internal hip rotation higher than 35 degrees and symptoms that don't pass the knee.

Exclusion Criteria:

* subjects presenting symptoms that pass the knee;
* impairment of neurologic signs like sensibility, muscle force and deep tendon reflex;
* a prior history of spondylolisthesis, spinal stenosis, inflammatory disease, cancer, musculoskeletal degenerative disease, pregnancy, disease and drugs that impairment the balance;
* subjects who received a HVLA manipulation of the lumbar spine at least three months earlier;
* will be excluded women older than 50 years, that don't will present a bone mineral density exam.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
pressure pain threshold assessment (algometer) | Within one day
  An algometer will used to assess the pressure pain threshold at baseline and following the intervention

SECONDARY OUTCOMES:
Clinical Prediction Rule | Within one day
  Variables which encompass the clinical prediction rule: symptoms lower than 16 days, Fear Avoidance-Beliefs Questionnaire lower than 19 in the work subscale, segmental lumbar hypermobility test in prone decubitus, internal hip rotation higher than 35 degrees and symptoms that don't pass the knee.
Center of pressure displacement | Within one day
  A force platform will be used to measure the displacement of the center of pressure (COP) in the anterior-posterior direction at baseline and following the intervention
Subjective pain assessment | Within one day
  Visual-analogue scale will be used to obtain a subjective assessment of pain at baseline and following the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jefferson F Loss, Phd, Study Director — Federal University of Rio Grande do Sul
Locations (1):
- Universidade Federal do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Fagundes Loss J, de Souza da Silva L, Ferreira Miranda I, Groisman S, Santiago Wagner Neto E, Souza C, Tarrago Candotti C. Immediate effects of a lumbar spine manipulation on pain sensitivity and postural control in individuals with nonspecific low back pain: a randomized controlled trial. Chiropr Man Therap. 2020 Jun 3;28(1):25. doi: 10.1186/s12998-020-00316-7. PMID 32487243